CLINICAL TRIAL: NCT06617156
Title: Comparison of Different Ventilator Measurement Methods of Rapid Shallow Breathing Index With Traditional Methods For Prediction Successful Extubation
Brief Title: Comparison of Ventilator Versus Traditional Measurement Methods of Rapid Shallow Breathing Index for Predicting Extubation Success
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202407034RIND
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Failure
Keywords: Ventilator weaning; Spirometry; Rapid shallow breathing index; Ventilator; Wright spirometer
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: RSBI Value Acquisition: All patients will undergo four methods to obtain the RSBI value Measurement Procedure: (1) The method of priority for measurement will be determined by random sampling (by drawing from an opaque envelope). (2) After each measurement, settings will return to baseline, and the next measurement can only occur after 10 minutes. (3) Collecting Ventilation Data: After changing the ventilation mode, wait 2 minutes to ensure stable breathing, then divide MV by RR to obtain tidal volume, and use RR divided by VT to obtain the RSBI value. (4)Simultaneous Measurement of EELI Changes Using Four Methods with EIT
  Interventions: Other: RSBI Value Evaluation

INTERVENTIONS:
Other: RSBI Value Evaluation — Spirometer Measurement: The traditional method for calculating RSBI involves the use of a spirometer (Wright MK20; Ferraris Medical Ltd., Hertford, England), equipped with a disposable bacterial filter at the front end, connected to the artificial airway to measure the minute ventilation of the patient's spontaneous breathing over one minute.
  Three Measurement Methods from the Ventilator: A. PSV at 5 cmH2O with PEEP at 5 cmH2O B. CPAP at 5 cmH2O C. CPAP at 0 cmH2O.
  Electrical impedance tomography (EIT) will be secured around the patient's thorax using a silicone belt, positioned at the fifth or sixth intercostal space, with 16 evenly spaced electrodes. Measurement data will be obtained by passing a small electrical current around the chest, utilizing the principle of resistance.

SUMMARY:
The Rapid Shallow Breathing Index (RSBI) (respiratory rate f / tidal volume VT) is a crucial indicator for predicting whether a patient can successfully wean off mechanical ventilation.

This study aims to explore the clinical value of measuring RSBI using different methods in predicting successful extubation. Study Methods: A prospective study was conducted in the medical and surgical intensive care units of a teaching hospital. Data were collected from patients who required intubation and mechanical ventilation due to respiratory failure from August 2024 to July 2026. The RSBI measured under different ventilator settings was compared with the traditional standard hand-held Wright spirometer measurement. The ventilator measurement methods were divided into three categories: PSV 5 cmH2O with PEEP 5 cmH2O, CPAP 5 cmH2O, and CPAP 0 cmH2O. The study analyzed the differences in RSBI measurements obtained by these methods and their ability to predict successful extubation, as well as other related factors, including the influence of different ventilator models, ventilation modes, and parameter settings on RSBI values. RSBI can vary across different patient populations and measurement methods. This study aims to validate the RSBI displayed by ventilators against the traditional standard measurement, providing a reliable predictive capability for successful extubation.

Furthermore, it seeks to facilitate clinical application and assist healthcare providers in determining the appropriate timing for extubation, reducing unnecessary prolonged use or premature removal of mechanical ventilation, and thereby lowering the incidence of complications and healthcare costs.

DETAILED DESCRIPTION:
In the Intensive Care Unit (ICU), approximately 25% of patients undergoing mechanical ventilation may experience difficulties during weaning from the ventilator. This can lead to delayed extubation, prolonged mechanical ventilation, increased length of stay in the hospital or ICU, and higher healthcare costs. On the other hand, premature extubation can result in secondary complications, increasing morbidity and mortality rates in the ICU. About 15% of patients who stop mechanical ventilation require reintubation within 48 hours. Therefore, it is crucial for intensivists to determine the appropriate timing for weaning from mechanical ventilation and successful extubation.

A study by Yang and Tobin in 1991 discovered that the ratio of respiratory rate to tidal volume (f/VT), known as the Rapid Shallow Breathing Index (RSBI), can serve as a predictor for successful weaning from mechanical ventilation. An RSBI value of <105 is considered indicative of a higher likelihood of successful extubation, while an RSBI value of >105 suggests a greater chance of weaning failure. The Wright spirometer is commonly used in clinical practice to measure RSBI. In practice, the spirometer is connected to the artificial airway, and the ventilator is disconnected for a 60-second respiratory measurement, without the need for additional complex equipment.

However, due to advancements in medical technology, ventilator parameters can also be used to calculate RSBI during Spontaneous Breathing Trials (SBT). Utilizing the ventilator to assess RSBI avoids interruptions in ventilation and reduces measurement risks. Research has shown that ventilator-calculated RSBI is convenient for clinical use and is feasible in predicting weaning outcomes. Nevertheless, variations in ventilator models, such as differences in base flow, type of ventilator, pressure compensation, Positive End-Expiratory Pressure (PEEP), and bias flow, may affect the accuracy of RSBI measurements obtained from the ventilator.

This study aims to further explore whether different measurement methods affect the accuracy of RSBI. However, weaning profiles should be evaluated comprehensively using additional parameters beyond RSBI, especially for patients requiring airway protection, increased secretions, or poor cough strength. Factors such as cough strength and the amount of secretions should be considered. A study on Chronic Obstructive Pulmonary Disease (COPD) patients found that early RSBI measurements did not accurately predict success in SBT; thus, this study will also analyze different disease diagnoses to provide reference for clinical assessment.

End-expiratory lung volume (EELV) is the lung volume at the end of expiration, representing the balance point between chest wall elastic recoil and lung collapse tendency, and is a major factor in determining lung oxygenation capacity. Changes in EELV are clinically significant, with studies indicating that a decrease in dorsal EELV slope is a strong predictor of lung collapse. Additionally, changes in EELV during SBT may be related to the patient's ability to successfully wean from mechanical ventilation. Electrical Impedance Tomography (EIT) measures changes in lung impedance based on variations in tissue and air distribution, providing cross-sectional images. EELV can be estimated from End-expiratory Lung Impedance (EELI), which will be included as an analysis parameter alongside different RSBI measurement methods.

Hypothesis: There is no significant difference between RSBI values obtained from ventilator measurements and those obtained using traditional handheld spirometry in predicting successful extubation.

Clinical Benefits: Traditional handheld spirometry requires temporarily disconnecting the ventilator, exposing staff to aerosolized droplets and potentially causing hypoxemia in patients dependent on oxygen support, which may lead to abnormal physiological parameters and increased patient risk. During the COVID-19 pandemic, traditional spirometry was not suitable due to airborne infection control requirements, and concerns about cross-infection between patients with reusable Wright spirometers were significant. Using the ventilator to measure RSBI is a feasible alternative. Currently, SBT is commonly used to evaluate extubation success in critically ill patients. Using the ventilator for RSBI measurements during SBT facilitates data acquisition and reduces environmental contamination between the ventilator and the patient.

There is still debate over the standard value for RSBI measurements obtained from ventilators compared to traditional methods. Some studies indicate similar results between traditional spirometry and ventilator-measured RSBI, while others show significantly higher RSBI values with traditional spirometry. This study will compare three different ventilator measurement methods with traditional standard measurements to explore differences in predicting extubation success. Additionally, changes in EELI will be compared across the four RSBI measurement methods.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Admission to the Intensive Care Unit (ICU).
* Endotracheal intubation with mechanical ventilation for more than 24 hours.
* P/F ratio > 150; FiO2 ≤ 40% and Positive End-Expiratory Pressure (PEEP) ≤ 8 cmH2O.
* Hemodynamically stable, without the need for vasoactive drugs or requiring only low doses.

Exclusion Criteria:

* Significant cardiac ischemia or arrhythmia.
* Patients with a tracheostomy.
* Patients with an endotracheal tube with an internal diameter smaller than 7.0 mm.
* Patients who have undergone repeated intubations within the past month.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients for whom the attending physician anticipates initiation of a Spontaneous Breathing Trial (SBT) and plans for extubation.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-16 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
RSBI Measured by the Ventilator | 60 minutes
  Accuracy of Predicting Extubation Success Using RSBI Measured by the Ventilator

SECONDARY OUTCOMES:
bias flow settings within different ventilators influence RSBI measurements. | 60 minutes
  Comparison of the Impact of Different Ventilator Bias Flows on RSBI Values: Analyze how variations in bias flow settings within different ventilators influence RSBI measurements.
Comparison of RSBI Values with and without PEEP in COPD Patients | 60 minutes
  Comparison of RSBI Values with and without PEEP in COPD Patients: Assess differences in RSBI values for Chronic Obstructive Pulmonary Disease (COPD) patients with and without the application of PEEP.
End-Expiratory Lung Impedance (EELI) Measured | 60 minutes
  Comparison of End-Expiratory Lung Impedance (EELI) Measured by Electrical Impedance Tomography (EIT) Across Four Measurement Methods: Use EIT to compare EELI measurements obtained from four different RSBI measurement methods.
Different Ventilator Inspiratory Pressures (PS) and Expiratory Pressures (PEEP) | 60 minutes
  Comparison of RSBI Values and Predictive Capability Based on Different Ventilator Inspiratory Pressures (PS) and Expiratory Pressures (PEEP): Evaluate how variations in inspiratory pressure (PS) and expiratory pressure (PEEP) affect RSBI values and their predictive accuracy for extubation success.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ramirez-Torres CA, Rivera-Sanz F, Sufrate-Sorzano T, Pedraz-Marcos A, Santolalla-Arnedo I. Closed Endotracheal Suction Systems for COVID-19: Rapid Review. Interact J Med Res. 2023 Jan 10;12:e42549. doi: 10.2196/42549. PMID 36548950
- [Result] Kheir F, Myers L, Desai NR, Simeone F. The effect of flow trigger on rapid shallow breathing index measured through the ventilator. J Intensive Care Med. 2015 Feb;30(2):103-6. doi: 10.1177/0885066613504538. Epub 2013 Sep 24. PMID 24067546
- [Result] Souza LC, Lugon JR. The rapid shallow breathing index as a predictor of successful mechanical ventilation weaning: clinical utility when calculated from ventilator data. J Bras Pneumol. 2015 Nov-Dec;41(6):530-5. doi: 10.1590/S1806-37132015000000077. PMID 26785962
- [Result] Patel KN, Ganatra KD, Bates JH, Young MP. Variation in the rapid shallow breathing index associated with common measurement techniques and conditions. Respir Care. 2009 Nov;54(11):1462-6. PMID 19863829
- [Result] Desai NR, Myers L, Simeone F. Comparison of 3 different methods used to measure the rapid shallow breathing index. J Crit Care. 2012 Aug;27(4):418.e1-6. doi: 10.1016/j.jcrc.2011.07.070. Epub 2011 Sep 29. PMID 21958982
- [Result] Duarte H, Fran A DLG, Portes MCF, Faria APAJ, Fontes RM, Wittmer VNLO, Barbalho-Moulim MC, Paro FVM. Comparison of different methods of obtaining the rapid shallow breathing index. Braz J Anesthesiol. 2023 Sep-Oct;73(5):578-583. doi: 10.1016/j.bjane.2021.05.001. Epub 2021 May 15. PMID 34004236
- [Result] Dasta JF, McLaughlin TP, Mody SH, Piech CT. Daily cost of an intensive care unit day: the contribution of mechanical ventilation. Crit Care Med. 2005 Jun;33(6):1266-71. doi: 10.1097/01.ccm.0000164543.14619.00. PMID 15942342
- [Result] Esteban A, Ferguson ND, Meade MO, Frutos-Vivar F, Apezteguia C, Brochard L, Raymondos K, Nin N, Hurtado J, Tomicic V, Gonzalez M, Elizalde J, Nightingale P, Abroug F, Pelosi P, Arabi Y, Moreno R, Jibaja M, D'Empaire G, Sandi F, Matamis D, Montanez AM, Anzueto A; VENTILA Group. Evolution of mechanical ventilation in response to clinical research. Am J Respir Crit Care Med. 2008 Jan 15;177(2):170-7. doi: 10.1164/rccm.200706-893OC. Epub 2007 Oct 25. PMID 17962636
- [Result] Goncalves EC, Lago AF, Silva EC, de Almeida MB, Basile-Filho A, Gastaldi AC. How Mechanical Ventilation Measurement, Cutoff and Duration Affect Rapid Shallow Breathing Index Accuracy: A Randomized Trial. J Clin Med Res. 2017 Apr;9(4):289-296. doi: 10.14740/jocmr2856w. Epub 2017 Feb 21. PMID 28270888
- [Result] Vetrugno L, Guadagnin GM, Brussa A, Orso D, Garofalo E, Bruni A, Longhini F, Bove T. Mechanical ventilation weaning issues can be counted on the fingers of just one hand: part 1. Ultrasound J. 2020 Mar 13;12(1):9. doi: 10.1186/s13089-020-00161-y. PMID 32166566
- [Result] Coplin WM, Pierson DJ, Cooley KD, Newell DW, Rubenfeld GD. Implications of extubation delay in brain-injured patients meeting standard weaning criteria. Am J Respir Crit Care Med. 2000 May;161(5):1530-6. doi: 10.1164/ajrccm.161.5.9905102. PMID 10806150
- [Result] McConville JF, Kress JP. Weaning patients from the ventilator. N Engl J Med. 2012 Dec 6;367(23):2233-9. doi: 10.1056/NEJMra1203367. No abstract available. PMID 23215559
- [Result] Yang KL, Tobin MJ. A prospective study of indexes predicting the outcome of trials of weaning from mechanical ventilation. N Engl J Med. 1991 May 23;324(21):1445-50. doi: 10.1056/NEJM199105233242101. PMID 2023603
- [Result] Meade M, Guyatt G, Cook D, Griffith L, Sinuff T, Kergl C, Mancebo J, Esteban A, Epstein S. Predicting success in weaning from mechanical ventilation. Chest. 2001 Dec;120(6 Suppl):400S-24S. doi: 10.1378/chest.120.6_suppl.400s. PMID 11742961
- [Result] Rittayamai N, Ratchaneewong N, Tanomsina P, Kongla W. Validation of rapid shallow breathing index displayed by the ventilator compared to the standard technique in patients with readiness for weaning. BMC Pulm Med. 2021 Oct 2;21(1):310. doi: 10.1186/s12890-021-01680-7. PMID 34600522
- [Result] Schmidt GA, Girard TD, Kress JP, Morris PE, Ouellette DR, Alhazzani W, Burns SM, Epstein SK, Esteban A, Fan E, Ferrer M, Fraser GL, Gong MN, L Hough C, Mehta S, Nanchal R, Patel S, Pawlik AJ, Schweickert WD, Sessler CN, Strom T, Wilson KC, Truwit JD; ATS/CHEST Ad Hoc Committee on Liberation from Mechanical Ventilation in Adults. Official Executive Summary of an American Thoracic Society/American College of Chest Physicians Clinical Practice Guideline: Liberation from Mechanical Ventilation in Critically Ill Adults. Am J Respir Crit Care Med. 2017 Jan 1;195(1):115-119. doi: 10.1164/rccm.201610-2076ST. PMID 27762608
- [Result] Na SJ, Ko RE, Nam J, Ko MG, Jeon K. Comparison between pressure support ventilation and T-piece in spontaneous breathing trials. Respir Res. 2022 Feb 7;23(1):22. doi: 10.1186/s12931-022-01942-w. PMID 35130914
- [Result] Karthika M, Al Enezi FA, Pillai LV, Arabi YM. Rapid shallow breathing index. Ann Thorac Med. 2016 Jul-Sep;11(3):167-76. doi: 10.4103/1817-1737.176876. PMID 27512505
- [Result] Purro A, Appendini L, De Gaetano A, Gudjonsdottir M, Donner CF, Rossi A. Physiologic determinants of ventilator dependence in long-term mechanically ventilated patients. Am J Respir Crit Care Med. 2000 Apr;161(4 Pt 1):1115-23. doi: 10.1164/ajrccm.161.4.9812160. PMID 10764299
- [Result] Cheng JC, Chen HC, Jerng JS, Kuo PH, Wu HD. End-Expiratory Lung Volumes During Spontaneous Breathing Trials in Tracheostomized Subjects on Prolonged Mechanical Ventilation. Respir Care. 2021 Nov;66(11):1704-1712. doi: 10.4187/respcare.08957. Epub 2021 Aug 31. PMID 34465570
- See also: Sermkaew T, Kongpolprom N. Electrical impedance tomography monitoring for predicting lung collapse after positive end expiratory pressure decrement in recovering acute respiratory distress syndrome. European Respiratory Journal. 2021;58. — http://erj.ersjournals.com/content/58/suppl_65/OA4023